CLINICAL TRIAL: NCT05813782
Title: The Effect of Baby Massage on Postpartum Depression and Maternal Attachment in the Postpartum Period: A Randomized Controlled Study
Brief Title: The Effect of Baby Massage on Postpartum Depression and Maternal Attachment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayla KORKMAZ, asst. prof., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-KAEK-084
Record Dates: First submitted 2023-03-23; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Depression, Postpartum; Maternal Behavior; Attachment
Keywords: Primiparous mother; Baby massage; Postpartum depression; Maternal attachment
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention arms (No Intervention): Primiparous mothers in this group answered the postpartum depression scale (pre-test) before discharge from the hospital. No intervention was made in addition to routine postnatal care. Primiparous mothers answered the maternal attachment scale and the postpartum depression scale (post-test) on postpartum 42nd day.
- Experimental arms (Experimental): Primiparous mothers in the experimental group answered the postpartum depression scale before baby massage training. Afterwards, baby massage training (30 min.) was given. Baby model, baby massage video CD and brochure were used in the training. Primiparous mothers were told to apply baby massage regularly for 15 minutes, once a day, every day from the 5th to 42nd day after birth. An "Baby Massage Follow-up Form" was given to primiparous mothers to record the days of massage. Baby massage application order was provided by phone calls twice a week. Primiparous mothers answered the maternal attachment scale and the postpartum depression scale (post-test) on postpartum 42nd day.
  Interventions: Behavioral: Baby Massage

INTERVENTIONS:
Behavioral: Baby Massage — Baby massage training (30 minutes) was given to primiparous mothers before they were discharged from the hospital. Baby massage training consists of sections that explain the importance of massage, preparation for massage, stages of baby massage and situations that need attention. Primiparous mothers were told to do this massage to their babies in the postpartum period. Baby massage video CD, brochure and baby oil were given to primiparous mothers for an effective baby massage.
  Arms: Experimental arms

SUMMARY:
This study was conducted to determine the effect of baby massage on postpartum depression and maternal attachment in the postpartum period.

DETAILED DESCRIPTION:
The transition to motherhood is one of the life stages that brings about stress and change. Primiparous mothers, who will experience motherhood for the first time due to anxiety about the unknown, may experience more stress and their communication with their babies may deteriorate. In this process, the mother's seeing, touching and interacting with her baby positively affects her perception of her baby. The easiest and most natural way to do this is baby massage. Touching and massaging the baby maintains the baby's body contact, which strengthens the baby's sense of trust and supports the mother's development of attachment behavior. It also reduces mothers' levels of stress hormones such as cortisol and relieves depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous,
* Cesarean section,
* Having a single baby,
* Between the ages of 19-35,
* Literate
* Effective communication.

Exclusion Criteria:

* Having a premature baby,
* Mother and baby have a disease that prevents massage,
* Loss of vision and hearing.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — focused on primiparous mothers
Enrollment: 90 (Estimated)
Dates: Start 2022-09-03 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Postpartum depression | Postpartum 42nd day
  The Edinburgh postpartum depression scale (EPDS) was used to determine the level of postpartum depression. EPDS is a 4-point Likert-type scale consisting of 10 questions and is scored between 0-3. The total score of the scale is obtained by summing the item scores. People with a score above 12 points are considered a risk group. The lowest score is 0 and the highest score is 30.
  Primiparous mothers answered before training (pretest) and postpartum 42nd day (posttest).
Maternal attachment | Postpartum 42nd day
  The level of maternal attachment was assessed using the " The Maternal Attachment Inventory (MAI)". The inventory consists of 26 Likert type items. Each item is scored between 1 and 4. Therefore, the minimum score of the inventory is 26 and the maximum score is 104. A high score indicates high attachment to the mother.
  Primiparous mothers answered on postpartum 42nd day (posttest).

CONTACTS AND LOCATIONS:
Overall Officials: Ayla KORKMAZ, asst. prof., Principal Investigator — Tokat Gaziosmanpaşa University
Locations (1):
- Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No